CLINICAL TRIAL: NCT03593889
Title: Jockey Club JoyAge: Holistic Support Project for Elderly Mental Wellness
Brief Title: Collaborative Stepped Care and Peer Support Programme for Older People At-Risk of or With Depression
Acronym: JCJoyAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Caritas Medical Centre, Hong Kong (Other); Christian Family Service Centre (Other); Haven of Hope Hospital (Other); Hong Kong Sheng Kung Hui Lady MacLehose Centre (Unknown); The Mental Health Association of Hong Kong (Other); New Life Psychiatric Rehabilitation Association (Other)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EA1709021
Record Dates: First submitted 2018-05-29; First posted 2018-07-20 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Depressive Symptoms
Keywords: Collaborative stepped care; Peer support; Early identification; Selective prevention; Indicated prevention
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The intervention group will receive a collaborative stepped care programme provided by registered social workers and trained peer supporters from elderly or mental health service units (NGOs) according to level of risks, symptom severity, and intervention response. Home visits or other format of contact will be delivered by trained peer supporters employed by NGOs to detect and engage hidden cases.
  The control group will receive treatment as usual, which will be determined by the responsible worker from NGO units.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a collaborative stepped care programme provided by registered social workers and trained peer supporters from elderly or mental health service units (NGOs) according to level of risks, symptom severity, and intervention response. Home visits or other format of contact will be delivered by trained peer supporters employed by NGOs to detect and engage hidden cases.
  Interventions: Behavioral: Collaborative stepped care and peer support programme
- Control group (Other): The control group will receive treatment as usual, which will be determined by the responsible worker from NGO units.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Collaborative stepped care and peer support programme — For "at-risk" group, 4 weeks of "selective prevention" group sessions will be provided at the elderly service level by trained peer supporters with registered social worker supervision, on wellness topics tailored to the person's concern as entry point, packaged with mental health information, followed by a review.
  For mild group, 6-8 weeks of indicated prevention with psychoeducation or low-intensity psychotherapy would be provided. For moderate group, 6-8 weeks high-intensity cognitive behavioral therapy (CBT) would be provided. All intervention for depressed elderly would be conducted by registered social workers. The trained peer supporters will be matched to individual older adults to walk them through the process with regular follow-up for 1 year.
  Arms: Intervention group
Other: Treatment as usual — The control group will receive treatment as usual, which will be determined by the responsible workers from NGO units.
  Arms: Control group

SUMMARY:
To develop a viable and sustainable best practice model to promote elderly mental wellness and prevent elderly depression for Hong Kong, the Hong Kong Jockey Club Charities Trust has initiated a pilot holistic support project entitled "JC JoyAge: Holistic Support Project for Elderly Mental Wellness". Commenced in October 2016, this 3-year project will deliver six programmes: (1) social services staff training; (2) peer supporters certificate training; (3) outreach and engagement activities for at-risk older adults; (4) standardized prevention and early intervention service; (5) community education programmes; and (6) public awareness and public education activities in four pilot districts in Hong Kong, namely Kwun Tong, Sham Shui Po, Kwai Chung, and Tseung Kwan O. The project aims specifically to:

1. Evaluate the effectiveness of a collaborative stepped care and peer support programme in engaging older people at-risk of or with depression;
2. Evaluate the efficacy of the programme in reducing symptoms/risks and promoting wellbeing in older people at-risk of or with depression;
3. Investigate the impact of the programme on care resources utilization in these older adults.

DETAILED DESCRIPTION:
Elderly depression is a neglected problem affecting our entire society with grave consequences and high societal costs. Early intervention and prevention can be effective in addressing the problem. The challenges in implementing early intervention and prevention within the existing service platforms, however, are threefold: (1) fragmented services; (2) reactive services; and (3) stigma and low awareness. These challenges resulted in the current service overload and mismatch, which will be compounded by rapid population ageing and mental health workforce shrinkage. The study can address these challenges by (1) realigning existing mental health and elderly services; (2) productive ageing for outreach and engagement; and (3) building up capacity of a preventive network in the neighbourhood. This pilot project therefore combines models of collaborative stepped care and productive ageing, with systematic education programmes, to empower the neighbourhood in providing effective early intervention and prevention for elderly depression. In the four representative pilot districts of Kwun Tong, Sham Shui Po, Kwai Chung, and Tseung Kwan O, community mental health and elderly services will collaborate to deliver a stepped care service protocol for preventing and detecting elderly depression. In 3 years, this project will deliver six programmes: (1) social services staff training; (2) peer supporters certificate training; (3) outreach and engagement activities for at-risk older adults; (4) standardized prevention and early intervention service; (5) community education programmes; and (6) public awareness and public education activities. This will produce a mature service model tested in one-fifth of the districts in Hong Kong with different demographic and service characteristics; create a strong team of Peer Supporters and Social Workers in Elderly Mental Health with clinical competence in preventing elderly depression and promoting elderly mental wellness; significantly raise public and neighbourhood awareness and care for elderly mental wellness; reach out and serve 2,880 at-risk older adults and 960 depressed older adults; and provide evidence on the social impact of the model for further service rollout.

ELIGIBILITY:
Inclusion Criteria:

* residing in Kwun Tong, Kwai Chung, Tseung Kwan O, or Sham Shui Po; and
* have one or more known risk factor(s) for developing depression; and/or
* have depressive symptoms of mild level or above; and
* able to give informed consent to participate

Exclusion Criteria:

* known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia; and
* imminent suicidal risk; and
* difficulty in communication

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3702 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline depression at 12 months | Baseline and 12-month follow-up
  Depression will be measured by the Patient Health Questionnaire (PHQ-9). The total score will be used, ranging from 0 to 27. Higher scores indicate higher levels of depressive symptoms.

SECONDARY OUTCOMES:
Change from baseline loneliness at 12 months | Baseline and 12-month follow-up
  Loneliness will be measured by the UCLA loneliness scale (UCLA-3). The total score will be used, ranging from 0 to 9. Higher scores indicate greater loneliness.
Change from baseline life engagement at 12 months | Baseline and 12-month follow-up
  Life engagement will be assessed using the typical day interview - a semi-structured interview asking clients about their typical day activities
Change from baseline self-harm risk at 12 months | Baseline and 12-month follow-up
  Self-harm risk will be measured by the self-harm risk assessment checklist.
Change from baseline anxiety at 12 months | Baseline and 12-month follow-up
  Anxiety will be measured by the Generalized Anxiety Disorder scale (GAD-7). The total score will be used, ranging from 0 to 21. Higher scores indicate higher levels of anxiety symptoms.
Change from baseline cognitive function at 12 months | Baseline and 12-month follow-up
  Cognitive function will be measured by the Hong Kong Montreal Cognitive Assessment 5-Minute Protocol (HK-MoCA 5-Min). The total score will be used, ranging from 0 to 30. Higher scores indicate higher levels of cognitive function.
Change from baseline social capital at 12 months | Baseline and 12-month follow-up
  Participants will be asked to list out names of people who they would turn to when they feel down, and when they need help for trivial things.
Change from baseline health-related quality of life at 12 months | Baseline and 12-month follow-up
  Health-related quality of life will be measured by the EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L).
Change from baseline service utilization at 12 months | Baseline and 12-month follow-up
  Service utilization will be measured by the Client Service Receipt Inventory (CSRI).

CONTACTS AND LOCATIONS:
Overall Officials: Terry Lum, PhD, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong; Gloria Wong, PhD, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong
Locations (8):
- Hong Kong (8):
  - Hong Kong Sheng Kung Hui Lady MacLehose Centre, Kwai Chung
  - New Life Psychiatric Rehabilitation Association, Kwai Chung
  - Christian Family Service Centre, Kwun Tong
  - The Mental Health Association of Hong Kong, Kwun Tong
  - Caritas Hong Kong, Sham Shui Po
  - New Life Psychiatric Rehabilitation Association, Sham Shui Po
  - Christian Family Service Centre, Tseung Kwan O
  - Haven of Hope Christian Service, Tseung Kwan O

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong SMY, Leung DKY, Liu T, Ng ZLY, Wong GHY, Chan WC, Lum TYS. Comorbid anxiety, loneliness, and chronic pain as predictors of intervention outcomes for subclinical depressive symptoms in older adults: evidence from a large community-based study in Hong Kong. BMC Psychiatry. 2024 Nov 21;24(1):839. doi: 10.1186/s12888-024-06281-2. PMID 39574082
- [Derived] Liu T, Peng MM, Wong FHC, Leung DKY, Zhang W, Wong GHY, Lum TYS. Differential Associations Between Depressive Symptom-Domains With Anxiety, Loneliness, and Cognition in a Sample of Community Older Chinese Adults: A Multiple Indicators Multiple Causes Approach. Innov Aging. 2023 Jul 19;7(7):igad075. doi: 10.1093/geroni/igad075. eCollection 2023. PMID 37727600
- [Derived] Liu T, Leung DKY, Lu S, Kwok WW, Sze LCY, Tse SSK, Ng SM, Wong PWC, Lou VWQ, Tang JYM, Wong DFK, Chan WC, Kwok RYK, Lum TYS, Wong GHY. Collaborative community mental health and aged care services with peer support to prevent late-life depression: study protocol for a non-randomised controlled trial. Trials. 2022 Apr 11;23(1):280. doi: 10.1186/s13063-022-06122-1. PMID 35410292
- [Derived] Liu T, Lu S, Leung DKY, Sze LCY, Kwok WW, Tang JYM, Luo H, Lum TYS, Wong GHY. Adapting the UCLA 3-item loneliness scale for community-based depressive symptoms screening interview among older Chinese: a cross-sectional study. BMJ Open. 2020 Dec 10;10(12):e041921. doi: 10.1136/bmjopen-2020-041921. PMID 33303463

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03593889/Prot_SAP_002.pdf